CLINICAL TRIAL: NCT02392117
Title: A Multi-centre, Prospective, Non-interventional Study of Insulin Degludec Investigating the Safety and Effectiveness in a Real World Population With Type 1 and 2 Diabetes Mellitus
Brief Title: Investigating the Safety and Effectiveness of Insulin Degludec in a Real World Population With Type 1 and 2 Diabetes Mellitus
Acronym: ReFLeCT
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN1250-4189; U1111-1158-0248 (Other: WHO); ENCEPP/SDPP/7880 (Other: EU PAS)
Record Dates: First submitted 2015-03-12; First posted 2015-03-18 (Estimated); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — insulin degludec

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Insulin degludec
  Interventions: Drug: insulin degludec

INTERVENTIONS:
Drug: insulin degludec — Tresiba® will be prescribed by the physician under normal clinical practice conditions and will be obtained/ purchased from the chemist based on physician prescription. No treatment given.

SUMMARY:
This study is conducted in Europe. The aim of this non-interventional study is to investigate the safety and effectiveness of insulin degludec (Tresiba®) in a real world population with type 1 (T1DM) and 2 (T2DM) diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any study-related activities (Study-related activities are any procedure related to recording of data according to the protocol)
* Male or female patients at least 18 years of age at time of informed consent
* T1DM (diagnosed clinically) prior to inclusion in the study, and/or T2DM, insulin using patients (diagnosed clinically) prior to inclusion in the study
* Planned initiation with Tresiba®

Exclusion Criteria:

* Known or suspected hypersensitivity to Tresiba® or any of the excipients listed in Section 6.1 of the SmPC (Summary of Product Characteristics) or related products
* Previous participation in this study (i.e. provision of informed consent)
* Patients who have previously been treated with Tresiba®
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female patients aged at least 18 years of age with either T1DM or T2DM (insulin using) (clinically diagnosed) prior to visit 1, who signed an informed consent form, and whose physician plans to start Tresiba® treatment are eligible for entry in this study.
Sampling Method: Non-Probability Sample
Enrollment: 1262 (Actual)
Dates: Start 2015-03-16 (Actual); Primary Completion 2018-03-19 (Actual); Study Completion 2018-03-19 (Actual)

PRIMARY OUTCOMES:
Change in the number of any hypoglycaemic episodes | End of 4 week baseline period, end of 12 month observation period

SECONDARY OUTCOMES:
Change from baseline in HbA1c (glycosylated haemoglobin) | 0- 12 months
Change from baseline in FPG (Fasting Plasma Glucose) | 0-12 months
Change from the baseline period in the number of severe hypoglycaemic episodes | 0-12 months
Change from baseline in HR-QoL (health-related quality of life) questionnaire scores (PROs (patient reported outcome): SF-36 (short form 36), and DTSQ(Diabetes Treatment Satisfaction Questionnaire )) | 0-12 months

CONTACTS AND LOCATIONS:
Locations (8):
- Novo Nordisk Investigational Site, Aarhus, Denmark
- Novo Nordisk Investigational Site, München, Germany
- Novo Nordisk Investigational Site, Padua, Italy
- Novo Nordisk Investigational Site, Utrecht, Netherlands
- Novo Nordisk Investigational Site, Palma de Mallorca, Spain
- Novo Nordisk Investigational Site, Karlstad, Sweden
- Novo Nordisk Investigational Site, Zurich, Switzerland
- Novo Nordisk Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com

REFERENCES:
- [Result] Fadini GP, Feher M, Hansen TK, de Valk HW, Koefoed MM, Wolden M, Zimmermann E, Jendle J. Switching to Degludec From Other Basal Insulins Is Associated With Reduced Hypoglycemia Rates: A Prospective Study. J Clin Endocrinol Metab. 2019 Dec 1;104(12):5977-5990. doi: 10.1210/jc.2019-01021. PMID 31397845
- [Derived] Fadini GP, Giordano C, Salvi L, Nicolucci A; REFLECT Italian Study Group. Reduced Rates of Hypoglycemia in Type 1 or Type 2 Diabetes After Switching to Insulin Degludec: Results from the Italian Cohort of the ReFLeCT Study. Diabetes Ther. 2020 Dec;11(12):2909-2920. doi: 10.1007/s13300-020-00936-5. Epub 2020 Oct 3. PMID 33011923
- [Derived] de Valk HW, Feher M, Hansen TK, Jendle J, Koefoed MM, Rizi EP, Zimmermann E, Fadini GP. Switching to Degludec is Associated with Reduced Hypoglycaemia, Irrespective of Definition Used or Patient Characteristics: Secondary Analysis of the ReFLeCT Prospective, Observational Study. Diabetes Ther. 2020 Sep;11(9):2159-2167. doi: 10.1007/s13300-020-00875-1. Epub 2020 Jul 14. PMID 32666165
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com